CLINICAL TRIAL: NCT02826577
Title: Effects of Pregnenolone on Perceived Social Isolation: A Double-blind Randomized Electrical Neuroimaging Study
Brief Title: Effects of Pregnenolone on Perceived Social Isolation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left institution.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-0834
Record Dates: First submitted 2016-07-01; First posted 2016-07-11 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Perceived Social Isolation
MeSH Terms: interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pregnenolone 175mg (Active Comparator): - Single dose of 175mg
  Interventions: Drug: Pregnenolone 175mg
- Pregnenolone 400mg (Active Comparator): - Single dose of 400mg
  Interventions: Drug: Pregnenolone 400mg
- Placebo (Placebo Comparator): - Single dose of placebo
  Interventions: Drug: Placebo
- Matched healthy controls (No Intervention): - No intervention

INTERVENTIONS:
Drug: Pregnenolone 175mg — Single Dose 175mg
  Arms: Pregnenolone 175mg
Drug: Pregnenolone 400mg — Single Dose 400mg
  Arms: Pregnenolone 400mg
Drug: Placebo — Single Dose
  Arms: Placebo

SUMMARY:
No studies to date have examined the effects of pregnenolone on hypervigilance for social threat in individuals with perceived social isolation (PSI). We therefore are conducting a double-blind randomized research study combining three validated behavioral paradigms on social threat attention, perception of others, and emotion regulation with high-density electrical neuroimaging to probe the neuro-circuitry of social threat processing in young adults high in perceived social isolation two hours after the oral administration of 175mg pregnenolone (N = 24), 400mg of pregnenolone (N = 24), or placebo (N = 24). Such research has the potential to yield important insights into the neurobehavioral mechanisms of pregnenolone on hypervigilance for social threat and perception of others--- a first key step toward the development of adjunctive pregnenolone therapy in individuals with PSI.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80
* At least a score of 42 on the UCLA Loneliness scale.
* Right handed
* Normal or corrected eye sight

Exclusion Criteria:

* Medical history of cancer
* Steroid use
* Psychotropic drugs
* History of heart irregularities
* Have a counter indication to EEG
* Age <21 or >32
* Score less than 42 on UCLA loneliness scale
* Left handed
* Meet MINI criteria for anything but untreated major depressive disorder
* Uncorrected vision
* Current or past neurological disorder including epilepsy or traumatic brain injury
* Have a counter indication to electrical neuroimaging
* Under hormonal therapy (including, but not limited to, testosterone)
* Unstable mental illness
* History of bipolar disorder, schizophrenia, or psychotic disorder
* Current or recent (past 3 months) substance use or dependence
* Currently taking any medications that may have unfavorable interactions with pregnenolone

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cacioppo, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cacioppo S, Cacioppo JT. Why may allopregnanolone help alleviate loneliness? Med Hypotheses. 2015 Dec;85(6):947-52. doi: 10.1016/j.mehy.2015.09.004. Epub 2015 Sep 5. PMID 26365247
- [Background] Cacioppo S, Capitanio JP, Cacioppo JT. Toward a neurology of loneliness. Psychol Bull. 2014 Nov;140(6):1464-504. doi: 10.1037/a0037618. Epub 2014 Sep 15. PMID 25222636
- [Background] Pibiri F, Nelson M, Guidotti A, Costa E, Pinna G. Decreased corticolimbic allopregnanolone expression during social isolation enhances contextual fear: A model relevant for posttraumatic stress disorder. Proc Natl Acad Sci U S A. 2008 Apr 8;105(14):5567-72. doi: 10.1073/pnas.0801853105. Epub 2008 Apr 7. PMID 18391192
- [Background] Porcu P, O'Buckley TK, Leslie Morrow A, Adinoff B. Differential hypothalamic-pituitary-adrenal activation of the neuroactive steroids pregnenolone sulfate and deoxycorticosterone in healthy controls and alcohol-dependent subjects. Psychoneuroendocrinology. 2008 Feb;33(2):214-26. doi: 10.1016/j.psyneuen.2007.11.003. Epub 2007 Dec 21. PMID 18096321
- [Background] Rasmusson AM, Pinna G, Paliwal P, Weisman D, Gottschalk C, Charney D, Krystal J, Guidotti A. Decreased cerebrospinal fluid allopregnanolone levels in women with posttraumatic stress disorder. Biol Psychiatry. 2006 Oct 1;60(7):704-13. doi: 10.1016/j.biopsych.2006.03.026. Epub 2006 Aug 24. PMID 16934764
- [Background] Crowley SK, O'Buckley TK, Schiller CE, Stuebe A, Morrow AL, Girdler SS. Blunted neuroactive steroid and HPA axis responses to stress are associated with reduced sleep quality and negative affect in pregnancy: a pilot study. Psychopharmacology (Berl). 2016 Apr;233(7):1299-310. doi: 10.1007/s00213-016-4217-x. Epub 2016 Feb 9. PMID 26856852
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Marx CE, Keefe RS, Buchanan RW, Hamer RM, Kilts JD, Bradford DW, Strauss JL, Naylor JC, Payne VM, Lieberman JA, Savitz AJ, Leimone LA, Dunn L, Porcu P, Morrow AL, Shampine LJ. Proof-of-concept trial with the neurosteroid pregnenolone targeting cognitive and negative symptoms in schizophrenia. Neuropsychopharmacology. 2009 Jul;34(8):1885-903. doi: 10.1038/npp.2009.26. Epub 2009 Apr 1. PMID 19339966
- [Background] Pinna G, Costa E, Guidotti A. Fluoxetine and norfluoxetine stereospecifically and selectively increase brain neurosteroid content at doses that are inactive on 5-HT reuptake. Psychopharmacology (Berl). 2006 Jun;186(3):362-72. doi: 10.1007/s00213-005-0213-2. Epub 2006 Jan 24. PMID 16432684
- [Background] van Broekhoven F, Verkes RJ. Neurosteroids in depression: a review. Psychopharmacology (Berl). 2003 Jan;165(2):97-110. doi: 10.1007/s00213-002-1257-1. Epub 2002 Nov 6. PMID 12420152

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants started the trial and received the intervention.
Period: Overall Study
Arm/Group | Pregnenolone 175mg | Pregnenolone 400mg | Placebo | Matched Healthy Controls
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No data was collected or analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone 175mg | Pregnenolone 400mg | Placebo | Matched Healthy Controls | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous [unit: Participants]
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: EEG Results
Description: Evoked Brain Potentials (measured brain response that is the direct result of a specific cognitive event). Change from baseline EEG results at 8 weeks. Average the electrical brain activity evoked by each type of stimuli to calculate the evoked brain potentials (any stereotyped electrophysical response to a stimulus).
Time Frame: 8 weeks
Population: No data was collected or analyzed due to Principal Investigator leaving the institution.
Arm/Group | Pregnenolone 175mg | Pregnenolone 400mg | Placebo | Matched Healthy Controls
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Eye Movement Tracking
Description: Movements to first saccades. Change from baseline eye movement tracking results at 8 weeks.
Time Frame: 8 weeks
Population: No data was collected or analyzed due to Investigator leaving the institution.
Arm/Group | Pregnenolone 175mg | Pregnenolone 400mg | Placebo | Matched Healthy Controls
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Pregnenolone 175mg | Pregnenolone 400mg | Placebo | Matched Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT02826577/Prot_SAP_003.pdf
  • Informed Consent Form (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT02826577/ICF_001.pdf